CLINICAL TRIAL: NCT07349589
Title: A Randomized, Open-label, Single-dose, Parallel-design, Phase 1 Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetics of DW5524 in Healthy Adult Volunteers
Brief Title: Evaluate the Safety, Tolerability and Pharmacokinetics of DW5524 in Healthy Adult Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DW5524-101
Record Dates: First submitted 2026-01-07; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group1 (Experimental): Group1
  Interventions: Drug: DW5524
- Group2 (Experimental): Group2
  Interventions: Drug: DW5524
- Group3 (Experimental): Group3
  Interventions: Drug: DW5524
- Group4 (Experimental): Group4
  Interventions: Drug: DW5524-A

INTERVENTIONS:
Drug: DW5524 — DW5524
  Arms: Group1; Group2; Group3
Drug: DW5524-A — DW5524-A
  Arms: Group4

SUMMARY:
This study aimed to evaluate the safety and pharmacokinetic characteristics of DW5524 in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers aged 19 years or older at the time of screening
* Individuals weighing 50.0 kg or more and having a body mass index (BMI) between 18.0 kg/m2 and 30.0 kg/m2 at the time of screening

Exclusion Criteria:

* Those with a current or past medical history of clinically significant liver, kidney, nervous, mental, respiratory, endocrine, blood disease, tumor, genitourinary, cardiovascular, digestive, or musculoskeletal diseases.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
AUC0-t | up to 8 hour
  Pharmacodynamic DW5524
Cmax | up to 8 hour
  Pharmacodynamic DW5524

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, South Korea